CLINICAL TRIAL: NCT03392987
Title: A Single Arm, Open Label, Clinical Study of Cryopreserved Autologous CD34+ Cells Transduced with Lentiviral Vector Containing Human ARSA CDNA (OTL-200), for the Treatment of Early Onset Metachromatic Leukodystrophy (MLD)
Brief Title: A Safety and Efficacy Study of Cryopreserved OTL-200 for Treatment of Metachromatic Leukodystrophy (MLD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Orchard Therapeutics (Industry)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205756; 2017-001730-26 (EudraCT Number)
Record Dates: First submitted 2017-12-12; First posted 2018-01-08 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Lysosomal Storage Disease; Metachromatic Leukodystrophy
Keywords: OTL-200; Cryopreserved formulation; Gene therapy; Metachromatic leukodystrophy; MLD; Previously GSK2696274
MeSH Terms: conditions — Lysosomal Storage Diseases; Leukodystrophy, Metachromatic

STUDY DESIGN:
Intervention Model Description: This will be a single arm study. All subjects will receive OTL-200 gene therapy and will be followed up for 5 years post-gene therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OTL-200 gene therapy (Experimental): Eligible subjects will receive intravenous (IV) infusion of OTL-200 gene therapy. Subjects will also receive conditioning regimen with busulfan.
  Interventions: Genetic: OTL-200

INTERVENTIONS:
Genetic: OTL-200 — OTL-200 is an autologous CD34+ enriched cell fraction that contains CD34+ cells transduced with lentiviral vector that encodes for the human ARSA cDNA sequence
  Other Names: Previously GSK2696274

SUMMARY:
OTL-200 is autologous CD34+ cells transduced with lentiviral vector containing human arylsulfatase A (ARSA) complementary deoxyribonucleic acid (cDNA) used for the treatment of MLD. MLD is an autosomal recessive lysosomal storage disorder (LSD) characterized by severe and progressive demyelination affecting the central and peripheral nervous system. This study will assess safety and efficacy of treatment using cryopreserved formulation of OTL-200 in pediatric subjects with pre-symptomatic Early Onset MLD (Late Infantile (LI) to Early Juvenile (EJ) MLD) and early symptomatic EJ MLD.

ELIGIBILITY:
Inclusion Criteria:

* Documented biochemical and molecular diagnosis of MLD, based on ARSA activity below the normal range and identification of two disease-causing ARSA alleles, either known or novel mutations. Novel mutations will be analyzed with in silico prediction tools and excluded from being known common polymorphisms. In the case of a novel mutation(s), a 24-hour urine collection must show elevated sulfatide levels.
* Eligible subjects must have EITHER

  1. an older sibling affected by MLD (index case), whose age of symptom onset was <=6 years of age (i.e., had not celebrated 7th birthday). Subjects will be classified as LI, EJ or intermediate LI/EJ based on age of symptom onset in the index case and their ARSA genotype; LI: symptom onset in index case <=30 months of age and genotype typically 0/0; EJ: symptom onset in index case >30 months and <= 6 years of age with genotype typically 0/R; Intermediate LI/EJ: symptom onset in index case <= 6 years of age but unable to unambiguously characterize index case as LI or EJ OR
  2. if MLD is diagnosed in a pre-symptomatic child without an older affected sibling, (e.g.) incidentally or via newborn screening) and the totality of the data available to the investigator strongly suggest that the subject has an early onset variant of MLD likely to benefit from gene therapy, and the subject is <=6 years of age (i.e., has not celebrated 7th birthday), the subject may be considered eligible after discussion and approval by the Orchard medical monitor.
* Parental/guardian signed and dated informed consent.

Exclusion Criteria:

* If LI MLD variant, clinical manifestations of the disease defined as EITHER of the following:

  * delay in expected achievement of independent standing or independent walking, together with abnormal signs at neurological evaluation
  * Or documented neurological signs and symptoms of MLD associated with cognitive, motor, or behavioural functional impairment or regression (substantiated by neurological examination and/or neuropsychological tests appropriate for age).

If EJ MLD variant, symptoms of MLD resulting in the loss of capacity of walking independently as defined by a GMFC level ≥2 or symptoms consistent with cognitive impairment as defined by an IQ<85 using age-appropriate neurocognitive instruments.

NOTE: The following will not be exclusionary if present alone:

* Seizures
* Signs of the disease revealed at instrumental evaluations (Electroneurography [ENG] and brain MR)

  * Documented HIV infection (positive HIV RNA and/or anti-p24 antibodies).
  * Malignant neoplasia (except local skin cancer) or a documented history of hereditary cancer syndrome. Subjects with a prior successfully treated malignancy and a sufficient follow-up to exclude recurrence (based on oncologist opinion) can be included after discussion and approval by the Medical monitor.
  * Myelodysplasia, cytogenetic alterations characteristic of myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML), or other serious hematological disorders.
  * Subjects currently enrolled in other interventional trials.
  * Has previously undergone allogeneic hematopoietic stem cell transplantation and has evidence of residual cells of donor origin.
  * Previous gene therapy.
  * Has symptomatic herpes zoster, not responsive to specific treatment. Subjects with a recent history of herpes zoster may be included in the study. In such cases, inclusion, additional monitoring and treatment of the condition must be discussed and approved by the medical monitor.
  * Evidence of active tuberculosis (TB) based upon medical examination, chest imaging and TB testing i.e. QuantiFERON-TB Gold test and microbiological evidence. Subjects with latent tuberculosis, as documented by medical history and/or TB testing may be included in the study if receiving antibiotic prophylaxis (e.g. isoniazid). Inclusion, monitoring and treatment of TB in such subjects must be discussed and approved by the medical monitor.
  * Acute or chronic stable Hepatitis B as evidenced by positive Hepatitis B surface antigen (HBsAg) test result at screening or within 3 months prior to onset of conditioning and/or positive hepatitis B virus (HBV) DNA. Subjects with positive Hepatitis B core antibody due to prior resolved disease may be enrolled, only if a confirmatory negative Hepatitis B surface antigen and negative Hepatitis B DNA test are obtained. Inclusion, monitoring and treatment of hepatitis in such subjects must be discussed and approved by the medical monitor.
  * Presence of positive Hepatitis C RNA test result at screening; subjects who have previously tested positive for antibodies against hepatitis C can be treated, provided they demonstrate absence of ongoing infection using a nucleic acid test with a limit of quantification of <=15 international units/milliliter (IU/mL). Negative test results are required on at least 3 sequential occasions over a period of at least 4 weeks, after completion of treatment for hepatitis C, with the final test conducted no more than 3 days prior to cell harvest. Inclusion, monitoring and treatment of hepatitis in such subjects must be discussed and approved by the medical monitor.
  * End-organ dysfunction, severe active infection not responsive to treatment, or other severe disease or clinical condition which, in the judgment of the investigator, would make the subject inappropriate for entry into this study. In addition to the potential infections the PI should consider testing for other transmissible infectious agents listed in the European Union (EU) Cell and Tissue Directive as clinically appropriate and results discussed with the medical monitor prior to cell harvest.
  * Subjects with alanine transferase (ALT) >2x upper limit of normal (ULN) or total bilirubin >1.5xULN may be included only after discussed and agreed with the medical monitor and considered in the context of the criterion for excluding subjects with other severe disease.
  * Isolated elevation of total bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent of total.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure (GMFM) score | At 24 months post gene-therapy
  GMFM will evaluate subject's ability to perform specific tasks in different positions. The scoring range is between 100 percent and 0 percent, with 0 percent corresponding to loss of all voluntary movement.

SECONDARY OUTCOMES:
Change in Gross Motor Function Measure (GMFM) score | At 24 months and multiple visits up to 5 years post-gene therapy
  GMFM will evaluate subject's ability to perform specific tasks in different positions. The scoring range is between 100 percent and 0 percent, with 0 percent corresponding to loss of all voluntary movement.
Change in Gross Motor Function Classification (GMFC)-MLD score | At 24 months and multiple visits up to 5 years post-gene therapy
  GMFC-MLD will evaluate the change in motor function according to seven clinically relevant levels of walking, sitting, locomotion, trunk and head control. The scoring range is from 0 (walking without support with quality of performance normal for age) to 6 (loss of any locomotion as well as loss of any head and trunk control).
Change in neurological examinations | At 24 months and multiple visits up to 5 years post-gene therapy
  Neurological examinations will be performed to identify any signs and symptoms of MLD disease.
Change in Nerve Conduction Velocity (NCV) | At 24 months and multiple visits up to 5 years post-gene therapy
  NCV will be assessed by electroneurography which is a technique used to test and quantify the nerve conduction and impulse propagation along motor and sensory peripheral nerves.
Change in total score for brain magnetic resonance (MR) imaging | At 24 months and multiple visits up to 5 years post-gene therapy
  Brain MR will be assessed using modified Loes score where normal brain has a score of zero and increasing score reflects worsening disease and demyelination.
Change in neurocognitive function (Intelligence Quotient [IQ]) | At 24 months and multiple visits up to 5 years post-gene therapy
  Standardized, age-appropriate IQ tests will be administered.
Engraftment measured by percent Lentiviral (LV) positive clonogenic progenitors in bone marrow | At Day 30 and multiple visits up to 5 years post-gene therapy
  Engraftment of transduced cells will be determined by measuring the percentage of hematopoietic colony-forming cells harboring the integrated vector by quantitative polymerase chain reaction (qPCR).
Vector copy number (VCN) level in bone marrow mononuclear cells | At Day 30 and multiple visits up to 5 years post-gene therapy
  Engraftment of transduced cells will be determined by measuring the VCN per genome in bone marrow-derived cells.
VCN level in peripheral blood mononuclear cell (PBMCs) | At Day 60 and multiple visits up to 5 years post-gene therapy
  Engraftment of transduced cells will be determined by measuring the VCN per genome in PBMCs.
Change in Arylsulfatase A (ARSA) activity in total PBMCs | At Day 60 and multiple visits up to 5 years post-gene therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in circulating total PBMCs post-treatment.
Change in ARSA activity in PB CD15+ cells | At Day 60 and multiple visits up to 5 years post-gene therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in circulating CD15+ cells post-treatment.
Change in ARSA activity in PB CD14+ cells | At Day 60 and multiple visits up to 5 years post-gene therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in circulating CD14+ cells post-treatment.
Change in ARSA activity in cerebrospinal fluid (CSF) | At Day 90 and multiple visits up to 5 years post-gene therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in the Central Nervous System (CNS) post-treatment.
Safety and tolerability as measured by recording of adverse events (AEs), including conditioning regimen related toxicity and AEs, and non-conditioning related AEs | Up to 5 years post-gene therapy
  An AE is any untoward medical occurrence in a clinical study subjects, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as an serious adverse event (SAE).
Safety and tolerability as measured by number of subjects not achieving hematological recovery (i.e., engraftment failure) | By Day 60 post-gene therapy
  Hematological recovery will be defined as reconstitution of absolute neutrophil count (ANC ) > 500 neutrophils per microliter, associated with evidence of bone marrow recovery by Day 60.
Safety and tolerability as measured by incidences and titers of anti-ARSA antibodies | Up to 5 years post-gene therapy
  Serum samples will be collected for anti-ARSA antibody analysis.
Safety and tolerability as measured by absence of abnormal clonal proliferation (ACP) | Up to 5 years post gene-therapy
  Malignancy or ACP due to insertional oncogenesis will be evaluated using different tests and procedures.
Safety and tolerability as measured by absence of replication competent lentivirus (RCL) | baseline, 1, 3, 6, and 12 months, then once a year up to 5 years post gene-therapy
  Molecular monitoring of RCL will be carried out using an enzyme-linked immunosorbent assay (ELISA) test for serum human immunodeficiency virus (HIV) p24 antigen. A positive HIV p24 test result is subject to second level testing including: a) DNA PCR for vesicular stomatitis virus G (VSV-G) envelope (PBMC), and b) reverse transcription (RT)-PCR for serum HIV-pol ribonucleic acid (RNA) (plasma).

CONTACTS AND LOCATIONS:
Overall Officials: Orchard Clinical Trials, Study Director — Orchard Therapeutics
Locations (1):
- Ospedale San Raffaele - Telethon Institute for Gene Therapy (OSR-TIGET), Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fumagalli F, Calbi V, Gallo V, Zambon AA, Recupero S, Ciotti F, Sarzana M, Fraschini M, Scarparo S, De Mattia F, Miglietta S, Pierini C, Soncini M, Morena F, Montini E, Barzaghi F, Consiglieri G, Ferrua F, Migliavacca M, Tucci F, Fratini ES, Ippolito A, Silvani P, Calvi MR, Clerici A, Corti A, Facchini M, Locatelli S, Sangalli M, Zancan S, Miotto F, Natali Sora MG, Baldoli C, Martino S, Cordoba-Claros A, Moro SL, Gollop ND, Abate J, Yarzi MN, Nutkins P, Shenker A, Calissano M, Brooks J, Richardson A, Campbell L, Filippi M, Naldini L, Cicalese MP, Ciceri F, Bernardo ME, Aiuti A. Long-Term Effects of Atidarsagene Autotemcel for Metachromatic Leukodystrophy. N Engl J Med. 2025 Apr 24;392(16):1609-1620. doi: 10.1056/NEJMoa2405727. PMID 40267426